CLINICAL TRIAL: NCT00210990
Title: A Multicenter, Phase 3 Study of the Safety and Effectiveness of Doripenem in Complicated Lower Urinary Tract Infection or Pyelonephritis
Brief Title: Doripenem in the Treatment of Complicated Lower Urinary Tract Infection or Pyelonephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Peninsula Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005398
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Tract Infections; Pyelonephritis
Keywords: Complicated Urinary Tract Infections; Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — Doripenem

INTERVENTIONS:
Drug: doripenem

SUMMARY:
The purpose of this study is to assess the microbiological cure rate of doripenem in the treatment of patients with complicated urinary tract infection or pyelonephritis. The study will also characterize the safety and tolerability of treatment with doripenem in patients with complicated urinary tract infection or pyelonephritis.

DETAILED DESCRIPTION:
Doripenem is an antibiotic medication not yet approved by the US FDA. This is a phase 3, multi-center, prospective, open-label, single-arm study of doripenem in the treatment of complicated lower urinary tract infection or pyelonephritis in adults. Patients are hospitalized, but subsequently, patients may treated as outpatient or through home-based therapy at the discretion of the investigators. Conventional laboratory data will be collected from patients at specified times throughout the study. The primary endpoint is microbiological response measured at test of cure visit. The patients will receive doripenem with duration of therapy up to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complicated lower urinary tract infection or pyelonephritis

Exclusion Criteria:

* Women who are pregnant, nursing or of child-bearing potential and not using a medically accepted, effective method of birth control
* History of moderate or severe hypersensitivity reactions to antibiotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2004-03; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Microbiological response measured at test of cure visit at early follow-up.

SECONDARY OUTCOMES:
Clinical response (cure) assessed at early follow-up visit. Proportion of patients with sustained microbiological and clinical response measured at late follow-up visit. Safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Redman R, Damiao R, Kotey P, Kaniga K, Davies T, Naber KG. Safety and efficacy of intravenous doripenem for the treatment of complicated urinary tract infections and pyelonephritis. J Chemother. 2010 Dec;22(6):384-91. doi: 10.1179/joc.2010.22.6.384. PMID 21303745
- [Derived] Kaniga K, Flamm R, Tong SY, Lee M, Friedland I, Redman R. Worldwide experience with the use of doripenem against extended-spectrum-beta-lactamase-producing and ciprofloxacin-resistant Enterobacteriaceae: analysis of six phase 3 clinical studies. Antimicrob Agents Chemother. 2010 May;54(5):2119-24. doi: 10.1128/AAC.01450-09. Epub 2010 Mar 8. PMID 20211892
- [Derived] Zhanel GG, Ketter N, Rubinstein E, Friedland I, Redman R. Overview of seizure-inducing potential of doripenem. Drug Saf. 2009;32(9):709-16. doi: 10.2165/00002018-200932090-00001. PMID 19670912
- See also: A Multicenter, Phase 3 Study to Confirm the Safety and Efficacy of Intravenous Doripenem in Complicated Lower Urinary Tract Infection or Pyelonephritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=640&filename=CR005398_CSR.pdf